CLINICAL TRIAL: NCT07356726
Title: Finding My Way-UK: Promoting Positive Psychological Outcomes in People Living With and Beyond Curatively Treated Cancer: A Pilot Randomised Trial
Brief Title: Finding My Way-UK: Promoting Positive Psychological Outcomes in People Living With and Beyond Curatively Treated Cancer
Acronym: FMW-UK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edge Hill University (Other)
Collaborators: Flinders University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ETH2425-0268
Record Dates: First submitted 2025-12-08; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cancer Survivorship; Cancer; Neoplasms
Keywords: Cancer Survivorship; Benefit Finding; Psychosocial Intervention; Acceptability; Feasibility; Pilot Randomised Trial; Resilience; Hope; Subjective Well-Being; Curatively Treated; Online Intervention; Psycho-Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomised 1:1 to the Finding My Way-UK intervention or a treatment-as-usual control group, with both arms running concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Finding My Way-UK Intervention (Experimental): Participants receive immediate access to the Finding My Way-UK online psychosocial program for four weeks. The program includes six self-guided modules on topics such as: treatment and communication with treatment teams, coping with treatment side effects, managing emotions, identity and body image, social support, and post-treatment adjustment.
  Interventions: Behavioral: Finding My Way-UK
- Control - Information Pack (Other): Participants receive a digital information pack listing national psychological support resources for people living with and beyond cancer (e.g., Macmillan Cancer Support, Maggie's). This arm represents a treatment-as-usual control providing publicly available information but no structured psychosocial content.
  Interventions: Other: Treatment-As-Usual Control

INTERVENTIONS:
Behavioral: Finding My Way-UK — Self-guided, web-based psychosocial intervention integrating cognitive-behavioural, psychoeducational, and mindfulness-based strategies to support people living with and beyond curatively treated cancer. Six modules delivered online; participants complete flexibly over four weeks.
  Other Names: FMW-UK
  Arms: Finding My Way-UK Intervention
Other: Treatment-As-Usual Control — Digital information pack (PDF) signposting to existing UK cancer-support organisations and psychological resources. Distributed by email; no structured therapeutic program or study-specific content.
  Other Names: Information Pack Control
  Arms: Control - Information Pack

SUMMARY:
The goal of this pilot randomised trial is to evaluate whether an online psychosocial intervention (Finding My Way-UK) is feasible and acceptable for individuals living with and beyond curatively treated cancer. The main questions it aims to answer are:

1. Is Finding My Way-UK feasible and acceptable for individuals living with and beyond curatively treated cancer?
2. Are there preliminary signals of efficacy in benefit finding and other well-being outcomes (hope, resilience, and subjective well-being)?
3. What is the potential role of information-seeking styles and self-management self-efficacy?

Participants will be randomly assigned to one of two groups:

1. Finding My Way-UK Intervention group: access a four-week, self-guided online program with six modules covering coping with treatment side effects, managing emotions, social support, body image, and post-treatment adjustment.
2. Control group: receive a digital information pack listing national psychological support resources.

All study activities will take place online. Participants will complete questionnaires before the program, after four weeks, and three months later.

DETAILED DESCRIPTION:
Finding My Way-UK is a broad psychosocial intervention that integrates theoretical foundations from cognitive-behavioural therapy, psychoeducation, and exercises from third-wave approaches such as mindfulness meditation. Originally developed in Australia, the program demonstrated efficacy in reducing distress among women with breast cancer. It has since been culturally adapted for the UK cancer-care context and previously underwent a pilot trial assessing its applicability to UK participants and preliminary signals of efficacy on distress outcomes.

Based on feedback from that earlier trial, several design modifications have been introduced to enhance feasibility and engagement: (i) The intervention duration has been reduced from six weeks to four weeks; and (ii) Participants will have immediate access to all six modules upon logging in, rather than the previous sequential weekly release. Additionally, recruitment will be conducted entirely online through collaborations with cancer charities and social-media outreach.

To the best of our knowledge, this represents the first online, self-guided, broad psychosocial intervention that aims to assess positive psychological outcomes in individuals living with and beyond curatively treated cancer. This pilot trial is therefore intended to evaluate the feasibility and acceptability of the revised design and to provide preliminary data to inform a future, fully powered randomised controlled trial.

Benefit finding, hope, resilience, and subjective well-being will be assessed to explore preliminary signals of efficacy. Given the pilot nature of the study and the modest sample size, analyses of these outcomes will be descriptive and exploratory only, focusing on effect-size estimation and clinically meaningful change rather than formal hypothesis testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with any cancer within the past 12 months;
* Cancer is being (or, indeed, was) treated with curative intent;
* Aged 16 years or older;
* Possess sufficient English proficiency to provide informed consent and use the program;
* Able to access the internet and have access to an email address (or are willing to set an email address up with our help).

Exclusion Criteria:

* Diagnosis of cancer not being treated with curative intent (for example, metastatic, stage IV, or otherwise advanced-stage disease);
* And/Or have a severe comorbidity that may hinder their ability to participate fully (such as being unable to complete study procedures or provide informed consent).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | From enrolment of the first participant until the recruitment target is reached (up to 6 months)
  The feasibility of recruitment will be assessed by the number of participants enrolled in the study per month.
Intervention Adherence: Modules Accessed | At post-intervention (week 4)
  The level of engagement with the Finding My Way-UK program, defined as the number of intervention modules accessed (opened) by each participant on the Finding My Way-UK platform.
Intervention Adherence: Modules Completed | At post-intervention (week 4)
  The number of intervention modules completed by each participant on the Finding My Way-UK platform.
Retention Rate at Post-Intervention | At post-intervention (week 4)
  Assessed by the percentage of participants who complete the post-intervention outcome assessment.
Retention Rate at 3-Month Follow-Up | At 3 months post-intervention
  The percentage of participants who complete the 3-month post-intervention outcome assessment.
Qualitative Acceptability of the Intervention | At post-intervention (week 4)
  At baseline, participants will be asked an open-ended question about their expectations for the intervention, specifically what they hope will change or improve. At follow-up, participants will provide free-text responses describing any unexpected changes or impacts. Free-text responses will be subjected to basic thematic analysis to identify common themes relating to participant experience and acceptability.
Quantitative Acceptability of the Intervention | At post-intervention (week 4)
  At baseline, participants will be asked an open-ended question about their expectations for the intervention, specifically what they hope will change or improve. At follow-up, participants rate the extent to which the intervention met these expectations on a Likert scale ranging from 1 (not at all) to 10 (completely). Higher scores indicate greater acceptability.

SECONDARY OUTCOMES:
Change from Baseline in Benefit Finding Score | Baseline (pre-intervention), post-intervention (week 4), and 3 months post-intervention
  Measured using the Benefit Finding Scale (BFS). The BFS contains 17 items rated from 1 = not at all to 5 = extremely, summed to a total score range of 17-85, with higher scores indicating greater benefit finding. Analyses will be descriptive and exploratory, focusing on estimating pre-post effect sizes and the proportion of participants showing reliable improvement using Reliable Change Indices; no formal hypothesis testing will be performed.
Change from Baseline in Satisfaction with Life | Baseline (pre-intervention), post-intervention (week 4), and 3 months post-intervention
  Subjective well-being will be assessed with the Satisfaction with Life Scale (SWLS). The SWLS comprises 5 items rated from 1 = strongly disagree to 7 = strongly agree, summed to give a total score range of 5-35, where higher scores reflect greater life satisfaction.
Change from Baseline in Hope | Baseline (pre-intervention), post-intervention (week 4), and 3 months post-intervention
  Measured using the Herth Hope Index (HHI). The HHI includes 12 items rated 1 = strongly disagree to 4 = strongly agree, summed for a total score range of 12-48; higher values indicate greater hope.
Change from Baseline in Resilience | Baseline (pre-intervention), post-intervention (week 4), and 3 months post-intervention
  Measured using the Connor-Davidson Resilience Scale-10 (CD-RISC-10). Ten items rated 0 (not true at all) to 4 (true nearly all the time) yield a total score range of 0-40, with higher scores indicating greater resilience.

OTHER OUTCOMES:
Change from Baseline in Self-Management Self-Efficacy | Baseline (pre-intervention), post-intervention (week 4), and 3 months post-intervention
  Measured using the Self-Efficacy for Managing Chronic Disease Scale. Six items rated 1-10; mean score represents overall self-efficacy (higher scores indicate higher self-management self-efficacy).
Information-Seeking Style | At baseline (pre-intervention)
  Assessed using the Cancer Information-Seeking Preferences Questionnaire, a single-item measure that classifies participants into one of five information-seeking styles: intense seekers, complementary seekers, fortuitous seekers, minimal/uninterested seekers, or guarded avoiders.

CONTACTS AND LOCATIONS:
Overall Officials: Kian Hughes, PhD Candidate, Principal Investigator — Edge Hill University
Locations (1):
- Edge Hill University - Department of Psychology, Ormskirk, Lancashire, United Kingdom

REFERENCES:
- [Result] Loiselle CG. Cancer information-seeking preferences linked to distinct patient experiences and differential satisfaction with cancer care. Patient Educ Couns. 2019 Jun;102(6):1187-1193. doi: 10.1016/j.pec.2019.01.009. Epub 2019 Jan 18. PMID 30685191
- [Result] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Result] Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. J Trauma Stress. 2007 Dec;20(6):1019-28. doi: 10.1002/jts.20271. PMID 18157881
- [Result] Herth K. Abbreviated instrument to measure hope: development and psychometric evaluation. J Adv Nurs. 1992 Oct;17(10):1251-9. doi: 10.1111/j.1365-2648.1992.tb01843.x. PMID 1430629
- [Result] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Result] Hulbert-Williams NJ, Leslie M, Hulbert-Williams L, Koczwara B, Watson EK, Hall PS, Ashley L, Coulson NS, Jackson R, Millington S; Finding My Way UK Trial Steering Group; Beatty L. The Finding My Way UK Clinical Trial: Adaptation Report and Protocol for a Replication Randomized Controlled Efficacy Trial of a Web-Based Psychological Program to Support Cancer Survivors. JMIR Res Protoc. 2021 Sep 20;10(9):e31976. doi: 10.2196/31976. PMID 34542420
- [Result] Beatty L, Kemp E, Coll JR, Turner J, Butow P, Milne D, Yates P, Lambert S, Wootten A, Yip D, Koczwara B. Finding My Way: results of a multicentre RCT evaluating a web-based self-guided psychosocial intervention for newly diagnosed cancer survivors. Support Care Cancer. 2019 Jul;27(7):2533-2544. doi: 10.1007/s00520-018-4526-1. Epub 2018 Nov 9. PMID 30411239
- [Result] Beatty L, Koczwara B, Wade T. Evaluating the efficacy of a self-guided Web-based CBT intervention for reducing cancer-distress: a randomised controlled trial. Support Care Cancer. 2016 Mar;24(3):1043-51. doi: 10.1007/s00520-015-2867-6. Epub 2015 Aug 7. PMID 26248651
- [Result] Beatty L, Kemp E, Wade T, Koczwara B; Finding My Way study investigators. Finding My Way: protocol of a randomised controlled trial evaluating an internet self-help program for cancer-related distress. BMC Cancer. 2015 Apr 30;15:328. doi: 10.1186/s12885-015-1322-x. PMID 25924674
- [Result] Antoni MH, Lehman JM, Kilbourn KM, Boyers AE, Culver JL, Alferi SM, Yount SE, McGregor BA, Arena PL, Harris SD, Price AA, Carver CS. Cognitive-behavioral stress management intervention decreases the prevalence of depression and enhances benefit finding among women under treatment for early-stage breast cancer. Health Psychol. 2001 Jan;20(1):20-32. doi: 10.1037//0278-6133.20.1.20. PMID 11199062

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT07356726/Prot_SAP_000.pdf